CLINICAL TRIAL: NCT01097694
Title: A 28 Week, Treatment Randomized, Double -Blind, Placebo-controlled Study of the Effects of cKit Inhibition by Imatinib in Patients With Severe Refractory Asthma (KIA)
Brief Title: Effects of cKit Inhibition by Imatinib in Patients With Severe Refractory Asthma (KIA)
Acronym: KIA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Baim Institute for Clinical Research (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Elliot Israel, MD, Director of the Asthma Research Center, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2010P000170; U01HL102225 (NIH)
Record Dates: First submitted 2010-03-23; First posted 2010-04-02 (Estimated); Results first posted 2017-05-19 (Actual); Last update posted 2017-05-19 (Actual); Status verified 2017-05

CONDITIONS: Asthma
Keywords: cKIT inhibition in Asthma; Efficacy of Imatinib in severe resistent asthma.
MeSH Terms: conditions — Asthma | interventions — Imatinib Mesylate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Imatinib mesylate (Active Comparator): Group on active imatinib treatment
  Interventions: Drug: Imatinib mesylate
- Placebo (Placebo Comparator): Group on Placebo treatment
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Imatinib mesylate — Imatinib will be initiated at an oral dose of 200 mg (two 100 mg film-coated tables) per day during the first two weeks of treatment. If the treatment is well tolerated, an up-titration to 400 mg daily (four 100 mg film-coated tables) will occur.
  Other Names: Gleevec, Zoleta, Glivec, Ziatir
  Arms: Imatinib mesylate
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to see whether a new investigational drug (Imatinib) may help improve asthma in people whose symptoms are not well controlled with high dose inhaled corticosteroid treatment.

DETAILED DESCRIPTION:
Severe asthmatics remain poorly controlled despite high doses of standard asthma therapy or even daily doses of systemic corticosteroids or their equivalent. They account for a large proportion of the morbidity and mortality associated with asthma. Features that seem to characterize many patients with this disorder include persistent inflammation, symptoms, and airway hyperresponsiveness in the face of corticosteroid therapy. Mast cells are powerful, long-lived tissue dwelling effector cells that are resistant to corticosteroid effects and have been implicated in the pathobiology of asthma. Mast cells in the airway smooth muscle have been found to be the major distinguishing difference between asthmatic and non-asthmatic eosinophil airway disease; and putative circulating mast cell progenitors are increased 5 fold in asthma. Stem cell factor (SCF) is critical to mast cell homeostasis and upregulation and has pleiotropic effects on mast cells and eosinophils . SCF levels are elevated in relation to asthma severity and SCF antibodies block hyperresponsiveness and inflammation and remodeling in murine asthma models. Imatinib, a specific tyrosine kinase inhibitor, inhibits cKit (Kit), the receptor for SCF on mast cells. Imatinib at doses equivalent to, or below, doses safely used in humans, also mimics or exceeds anti-SCF effects in the murine asthma model. Therefore we would like to know Does imatinib, an inhibitor of Kit, ameliorate severe asthma, in association with effects on lung mast cell phenotype and/or function?

Specific Aims of the study are:

Specific Aim 1: To investigate whether, in patients with persistent airway responsiveness and poor asthma control despite intensive asthma therapy, 24 weeks of imatinib therapy results in a reduction in airway responsiveness and in secondary indicators of asthma control, airway inflammation, and structural changes in the airways.

Patients will be treated with imatinib in a randomized, double-blind, placebo controlled trial. Assessments will include methacholine and AMP reactivity, airway function, symptoms, airway wall thickness by CT scan, analysis of induced sputum, non-invasive markers of airway inflammation, and bronchoscopy including endobronchial biopsy and bronchoalveolar lavage - all before and at the end of therapy.

Specific Aim 2: To investigate whether, in patients with persistent airway responsiveness and poor asthma control despite intensive asthma therapy, 24 weeks of imatinib therapy results in changes in airway mast cell population and/or phenotype.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 18-65 years of age, diagnosed with asthma for at least 1 year;
2. Refractory asthma, defined as reporting that their asthma has not been completely controlled in the past 3 months despite continuous treatment with high-dose inhaled corticosteroids (ICS) and an additional controller medication, with or without continuous oral corticosteroids (OCS)

Exclusion Criteria:

1. Current smoking or smoking history of greater than 10 pack-years
2. Any other significant respiratory or cardiac disease, or the presence of clinically important comorbidities, including uncontrolled diabetes, uncontrolled coronary artery disease
3. If subject cannot undergo bronchoscopy procedure due to safety reasons
4. Previous treatment with Imatinib
5. A history of acute heart failure or chronic left sided heart failure
6. Uncontrolled systemic arterial hypertension
7. History of major bleeding or intracranial hemorrhage
8. History of immunodeficiency diseases, including HIV
9. Use of other investigational drugs at the time of enrollment, or within 30 days or 5 half-lives of enrollment, whichever is longer
10. History of malignancy of any organ system (other than localized basal cell carcinoma of the skin), treated or untreated, within the past 5 years, regardless of whether there is evidence of local recurrence or metastases.
11. Diagnosis of Hepatitis B or C.
12. History of alcohol abuse within 6 months of screening.
13. History of illicit drug abuse within 6 months of screening.
14. Regular use of anticoagulants (eg: Warfarin Sodium, Coumadin), amiodarone, carbamazepine, Cyclosporine, Rifampicin, or reverse transcriptase inhibitors

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2010-11; Primary Completion 2015-08 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elliot Israel, M.D, Principal Investigator — Brigham and Womens Hospital; Joshua Boyce, M.D, Principal Investigator — Brigham and Womens Hospital
Locations (7):
- United States (7):
  - University of Alabama, Birmingham, Alabama
  - Brigham and Womens Hospital, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - Columbia University, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Temple University, Philadelphia, Pennsylvania
  - University of Wisconsin, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Al-Muhsen SZ, Shablovsky G, Olivenstein R, Mazer B, Hamid Q. The expression of stem cell factor and c-kit receptor in human asthmatic airways. Clin Exp Allergy. 2004 Jun;34(6):911-6. doi: 10.1111/j.1365-2222.2004.01975.x. PMID 15196279
- [Background] Bischoff SC, Dahinden CA. c-kit ligand: a unique potentiator of mediator release by human lung mast cells. J Exp Med. 1992 Jan 1;175(1):237-44. doi: 10.1084/jem.175.1.237. PMID 1370529
- [Background] Brightling CE, Bradding P, Symon FA, Holgate ST, Wardlaw AJ, Pavord ID. Mast-cell infiltration of airway smooth muscle in asthma. N Engl J Med. 2002 May 30;346(22):1699-705. doi: 10.1056/NEJMoa012705. PMID 12037149
- [Background] Campbell E, Hogaboam C, Lincoln P, Lukacs NW. Stem cell factor-induced airway hyperreactivity in allergic and normal mice. Am J Pathol. 1999 Apr;154(4):1259-65. doi: 10.1016/S0002-9440(10)65377-1. PMID 10233863
- [Background] Carroll NG, Mutavdzic S, James AL. Increased mast cells and neutrophils in submucosal mucous glands and mucus plugging in patients with asthma. Thorax. 2002 Aug;57(8):677-82. doi: 10.1136/thorax.57.8.677. PMID 12149526
- [Background] Flood-Page P, Swenson C, Faiferman I, Matthews J, Williams M, Brannick L, Robinson D, Wenzel S, Busse W, Hansel TT, Barnes NC; International Mepolizumab Study Group. A study to evaluate safety and efficacy of mepolizumab in patients with moderate persistent asthma. Am J Respir Crit Care Med. 2007 Dec 1;176(11):1062-71. doi: 10.1164/rccm.200701-085OC. Epub 2007 Sep 13. PMID 17872493
- [Background] Proceedings of the ATS workshop on refractory asthma: current understanding, recommendations, and unanswered questions. American Thoracic Society. Am J Respir Crit Care Med. 2000 Dec;162(6):2341-51. doi: 10.1164/ajrccm.162.6.ats9-00. No abstract available. PMID 11112161
- [Background] Lukacs NW, Kunkel SL, Strieter RM, Evanoff HL, Kunkel RG, Key ML, Taub DD. The role of stem cell factor (c-kit ligand) and inflammatory cytokines in pulmonary mast cell activation. Blood. 1996 Mar 15;87(6):2262-8. PMID 8630386
- [Background] Nair P, Pizzichini MM, Kjarsgaard M, Inman MD, Efthimiadis A, Pizzichini E, Hargreave FE, O'Byrne PM. Mepolizumab for prednisone-dependent asthma with sputum eosinophilia. N Engl J Med. 2009 Mar 5;360(10):985-93. doi: 10.1056/NEJMoa0805435. PMID 19264687
- [Background] Reber L, Da Silva CA, Frossard N. Stem cell factor and its receptor c-Kit as targets for inflammatory diseases. Eur J Pharmacol. 2006 Mar 8;533(1-3):327-40. doi: 10.1016/j.ejphar.2005.12.067. Epub 2006 Feb 17. PMID 16483568
- [Background] Yuan Q, Austen KF, Friend DS, Heidtman M, Boyce JA. Human peripheral blood eosinophils express a functional c-kit receptor for stem cell factor that stimulates very late antigen 4 (VLA-4)-mediated cell adhesion to fibronectin and vascular cell adhesion molecule 1 (VCAM-1). J Exp Med. 1997 Jul 21;186(2):313-23. doi: 10.1084/jem.186.2.313. PMID 9221761
- [Derived] Cahill KN, Katz HR, Cui J, Lai J, Kazani S, Crosby-Thompson A, Garofalo D, Castro M, Jarjour N, DiMango E, Erzurum S, Trevor JL, Shenoy K, Chinchilli VM, Wechsler ME, Laidlaw TM, Boyce JA, Israel E. KIT Inhibition by Imatinib in Patients with Severe Refractory Asthma. N Engl J Med. 2017 May 18;376(20):1911-1920. doi: 10.1056/NEJMoa1613125. PMID 28514613

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from November 2010 until December 2014 in seven academic medical centers.
Pre-assignment Details: Following enrollment, 176 subjects entered a run-in period in which several inclusion criteria had to be met prior to randomization, including ACQ requirements and methacholine sensitivity, as well as safety and compliance requirements. 114 subjects who did not meet these inclusion criteria were not randomized.
Period: Overall Study
Arm/Group | Imatinib Mesylate | Placebo
Started | 32 | 30
Completed | 24 | 26
Not Completed | 8 | 4
Not completed — Adverse Event | 5 | 0
Not completed — Lost to Follow-up | 0 | 3
Not completed — Withdrawal by Subject | 3 | 1

BASELINE CHARACTERISTICS:
Population: severe asthmatics ages 18-65
Groups:
- Total: Total of all reporting groups
Arm/Group | Imatinib Mesylate | Placebo | Total
Number analyzed (Participants) | 32 | 30 | 62
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 32 | 30 | 62
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.2 (10.2) | 37.7 (11.8) | 40.1 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 18 | 37
  Male | 13 | 12 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 5 | 10
  Not Hispanic or Latino | 27 | 25 | 52
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 11 | 13 | 24
  White | 20 | 15 | 35
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 32 | 30 | 62

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean Methacholine Responsiveness as Assessed by the Provocation Concentration Causing a 20% Fall in Forced Expiratory Volume in One Second (FEV1) (PC20) at Month 3 and 6 Versus Baseline
Description: Our primary outcome was change in airway hyperresponsiveness, as assessed by PC20, from baseline to 3 and/or 6 months of therapy in imatinib treated participants as compared with controls. Change in PC20 was assessed using log2-transformed ratios of PC20 at month 3 and /or month 6 vs PC20 at baseline. Our null hypothesis was that the mean of this ratio will be 0 after log2-transformed. We used a linear mixed-effects model for a repeated-measures analysis to compare the primary outcome between the two groups.
  PC20 is determined by the provocation concentration of methacholine causing a 20% fall in forced expiratory volume in one second (FEV1).
Time Frame: Over 6 months from beginning of treatment
Measure: Mean (Standard Deviation); unit: Log2 Ratio
Arm/Group | Imatinib Mesylate | Placebo
Number analyzed (Participants) | 24 | 26
Log2 Ratio | 1.73 (0.52) | 1.07 (0.60)
Statistical Analysis 1: Comparison: Imatinib Mesylate vs Placebo; Our null hypothesis was that the mean of this ratio will be 0 after log2-transformed. The target enrollment was 60 assuming 10% drop-out for 54 completions which gave us 80% power to detect a doubling-dose change in PC20; Test type: Superiority; p < 0.05, Mixed Models Analysis

2. Secondary Outcome: Serum Total Tryptase
Description: Change in serum total tryptase after 24 weeks of imatinib vs placebo treatment
Time Frame: 6 months after start of treatment
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Imatinib Mesylate | Placebo
Number analyzed (Participants) | 19 | 23
ng/ml | -2.02 (2.32) | -0.56 (1.39)
Statistical Analysis 1: Comparison: Imatinib Mesylate vs Placebo; Test type: Superiority; p < 0.05, Regression, Linear; Adjusted for baseline

3. Secondary Outcome: Bronchoalveolar Lavage (BAL) Fluid Tryptase Level
Description: Change in BAL fluid tryptase levels after 24 weeks of imatinib vs. placebo
Time Frame: 6 months after start of treatment
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Imatinib Mesylate | Placebo
Number analyzed (Participants) | 21 | 26
ng/mL | -0.74 (2.35) | 0.43 (2.19)
Statistical Analysis 1: Comparison: Imatinib Mesylate vs Placebo; Test type: Superiority; p = 0.12, Regression, Linear; Adjusted for baseline

4. Secondary Outcome: Change in Maximum Post-Bronchodilator (BD) Forced Expiratory Volume in One Second (FEV1) %
Time Frame: 6 months after start of treatment
Measure: Mean (Standard Deviation); unit: % of predicted
Arm/Group | Imatinib Mesylate | Placebo
Number analyzed (Participants) | 24 | 26
% of predicted | 0.01 (0.2) | -0.08 (0.26)
Statistical Analysis 1: Comparison: Imatinib Mesylate vs Placebo; Test type: Superiority; p = 0.10, Regression, Linear; Adjusted for baseline

5. Secondary Outcome: Number of Asthma Exacerbations
Description: Number of asthma exacerbations experienced from randomization to study completion.
Time Frame: Up to 24 weeks
Measure: Number; unit: events
Arm/Group | Imatinib Mesylate | Placebo
Number analyzed (Participants) | 32 | 30
events | 16 | 20
Statistical Analysis 1: Comparison: Imatinib Mesylate vs Placebo; Test type: Superiority; p = 0.36, Poisson regression model

6. Secondary Outcome: FEV1 in Liters
Description: Change in FEV1 in treatment group compared to placebo group
Time Frame: 6 months after start of treatment
Measure: Mean (95% Confidence Interval); unit: L
Arm/Group | Imatinib Mesylate | Placebo
Number analyzed (Participants) | 32 | 30
L | 0.046 [0.036 to 0.056] | 0 [0 to 0]
Statistical Analysis 1: Comparison: Imatinib Mesylate vs Placebo; For FEV1 we used a linear mixed-effects model to assess the between-group difference in the change from baseline over weeks 8-24; Test type: Superiority; p < 0.05, Mixed Models Analysis; adjusted for baseline values

7. Secondary Outcome: FEV1%
Description: Change in FEV1% of predicted
Time Frame: 6 months after start of treatment
Measure: Mean (Standard Deviation); unit: % of predicted
Arm/Group | Imatinib Mesylate | Placebo
Number analyzed (Participants) | 24 | 27
% of predicted | 2.3 (8.86) | 0.78 (13.1)
Statistical Analysis 1: Comparison: Imatinib Mesylate vs Placebo; For FEV1% we used a linear mixed-effects model to assess the between-group difference in the change from baseline over weeks 8-24; Test type: Superiority; p = 0.06, Mixed Models Analysis; Adjusted for baseline

8. Secondary Outcome: Morning Peak Flow Measurement
Description: Change in patient-reported morning peak flow measurement (L/s)
Time Frame: 6 months after start of treatment
Measure: Mean (Standard Deviation); unit: L/second
Arm/Group | Imatinib Mesylate | Placebo
Number analyzed (Participants) | 19 | 20
L/second | 7.3 (46.1) | -6.4 (39.3)
Statistical Analysis 1: Comparison: Imatinib Mesylate vs Placebo; Test type: Superiority; p = 0.38, Mixed Models Analysis; Adjusted for baseline

9. Secondary Outcome: Evening Peak Flow
Description: Change in patient-reported evening peak flow measurement (L/s)
Time Frame: 6 months after start of treatment
Measure: Mean (Standard Deviation); unit: L/second
Arm/Group | Imatinib Mesylate | Placebo
Number analyzed (Participants) | 19 | 20
L/second | 8.3 (53.6) | -8.2 (37.2)
Statistical Analysis 1: Comparison: Imatinib Mesylate vs Placebo; Test type: Superiority; p = 0.31, Mixed Models Analysis; Adjusted for baseline

10. Secondary Outcome: Fractional Exhaled Nitric Oxide (FeNO)
Description: Change in Fractional Exhaled Nitric Oxide Measurement (ppb)
Time Frame: 6 months after start of treatment
Measure: Mean (Standard Deviation); unit: parts per billion
Arm/Group | Imatinib Mesylate | Placebo
Number analyzed (Participants) | 22 | 24
parts per billion | 7.89 (33.0) | -5.92 (33.2)
Statistical Analysis 1: Comparison: Imatinib Mesylate vs Placebo; Test type: Superiority; p = 0.11, Regression, Linear; Adjusted for baseline

11. Secondary Outcome: Asthma Control Questionnaire (ACQ)
Description: Change in patient-reported ACQ score The six-item Asthma Control Questionnaire (ACQ-6) is a scale from 0 to 6 with a lower value denoting an improvement in asthma control. The minimal important difference is 0.5.
Time Frame: 6 months after start of treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Imatinib Mesylate | Placebo
Number analyzed (Participants) | 24 | 27
units on a scale | -0.62 (0.96) | -0.49 (0.89)
Statistical Analysis 1: Comparison: Imatinib Mesylate vs Placebo; Test type: Superiority; p = 0.31, Regression, Linear; Adjusted for baseline

12. Secondary Outcome: Asthma Quality of Life Questionnaire (AQLQ)
Description: Change in patient-reported Asthma Quality of Life Questionnaire (AQLQ) score The asthma quality of life questionnaire (AQLQ) is a 32-item scale with a range from 1-7 with a higher value denoting improvement. The minimal important difference is 0.5.
Time Frame: 6 months after start of treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Imatinib Mesylate | Placebo
Number analyzed (Participants) | 20 | 24
units on a scale | 0.55 (1.0) | 0.25 (0.8)
Statistical Analysis 1: Comparison: Imatinib Mesylate vs Placebo; Test type: Superiority; p = 0.11, Regression, Linear; Adjusted for baseline

13. Secondary Outcome: Asthma Symptom Utility Index (ASUI)
Description: Change in patient reported ASUI score The asthma symptom utility index (ASUI) is a 10-item weighted scale with a range from 0.2 to 1 with a higher value indicating improvement. The minimal important difference is 0.09.
Time Frame: 6 months after start of treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Imatinib Mesylate | Placebo
Number analyzed (Participants) | 20 | 24
units on a scale | 0.07 (0.20) | 0.05 (0.18)
Statistical Analysis 1: Comparison: Imatinib Mesylate vs Placebo; Test type: Superiority; p = 0.62, Regression, Linear; Adjusted for baseline

14. Secondary Outcome: BAL Neutrophil %
Description: Change in BAL neutrophil percentage from baseline
Time Frame: 6 months after start of treatment
Measure: Mean (Standard Deviation); unit: % neutrophils
Arm/Group | Imatinib Mesylate | Placebo
Number analyzed (Participants) | 17 | 20
% neutrophils | -0.8 (5.6) | -0.4 (7.0)
Statistical Analysis 1: Comparison: Imatinib Mesylate vs Placebo; Test type: Superiority; p = 0.57, Regression, Linear; Adjusted for baseline

15. Secondary Outcome: BAL Eosinophil %
Description: Change in BAL eosinophil percentage
Time Frame: 6 months after start of treatment
Measure: Mean (Standard Deviation); unit: % eosinophils
Arm/Group | Imatinib Mesylate | Placebo
Number analyzed (Participants) | 17 | 26
% eosinophils | 2.55 (8.8) | -2.63 (10.4)
Statistical Analysis 1: Comparison: Imatinib Mesylate vs Placebo; Test type: Superiority; p = 0.15, Regression, Linear; Adjusted for baseline

16. Secondary Outcome: Bronchoalveolar Lavage (BAL) PGD2
Description: Change in bronchoalveolar lavage (BAL) PGD2 levels from baseline at 6 months
Time Frame: 6 months after start of treatment
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Imatinib Mesylate | Placebo
Number analyzed (Participants) | 21 | 26
pg/mL | 12.2 (57.2) | -4.2 (54.4)
Statistical Analysis 1: Comparison: Imatinib Mesylate vs Placebo; Test type: Superiority; p = 0.33, Regression, Linear; Adjusted for baseline

17. Secondary Outcome: Endobronchial Biopsy Total Tryptase-positive Mast Cells
Description: Change in endobronchial biopsy total tryptase-positive mast cells from baseline at 6 months
Time Frame: 6 months after start of treatment
Measure: Mean (Standard Deviation); unit: mast cells per mm2
Arm/Group | Imatinib Mesylate | Placebo
Number analyzed (Participants) | 23 | 26
mast cells per mm2 | -54.2 (96.5) | -32.3 (79.8)
Statistical Analysis 1: Comparison: Imatinib Mesylate vs Placebo; Test type: Superiority; p = 0.11, Regression, Linear; Adjusted for baseline

18. Secondary Outcome: Endobronchial Biopsy Smooth Muscle Tryptase-positive Mast Cells
Description: Change in the biopsy smooth muscle tryptase-positive mast cells from baseline at 6 months
Time Frame: 6 months after start of treatment
Measure: Mean (Standard Deviation); unit: mast cells per mm2
Arm/Group | Imatinib Mesylate | Placebo
Number analyzed (Participants) | 23 | 26
mast cells per mm2 | -102.7 (167.9) | -79.2 (157.3)
Statistical Analysis 1: Comparison: Imatinib Mesylate vs Placebo; Test type: Superiority; p = 0.07, Regression, Linear; Adjusted for baseline

19. Secondary Outcome: Blood Eosinophils
Description: Change in blood eosinophil count
Time Frame: 6 months after start of treatment
Measure: Mean (Standard Deviation); unit: eosinophils per microliter
Arm/Group | Imatinib Mesylate | Placebo
Number analyzed (Participants) | 20 | 20
eosinophils per microliter | -10.2 (50.6) | -2.6 (25.6)
Statistical Analysis 1: Comparison: Imatinib Mesylate vs Placebo; Test type: Superiority; p = 0.94, Regression, Linear; Adjusted for baseline

20. Secondary Outcome: Airway Wall Thickness
Description: Change in airway wall thickness as assessed by computerized tomography (CT)
Time Frame: 6 months after start of treatment
Measure: Mean (Standard Deviation); unit: % of airway
Arm/Group | Imatinib Mesylate | Placebo
Number analyzed (Participants) | 21 | 27
% of airway | -0.0040 (0.03) | -0.0027 (0.02)
Statistical Analysis 1: Comparison: Imatinib Mesylate vs Placebo; Test type: Superiority; p = 0.13, Regression, Linear; Adjusted for baseline

21. Secondary Outcome: Airway Wall Area
Description: Change in airway wall area as assessed by computerized tomography (CT)
Time Frame: 6 months after start of treatment
Measure: Mean (Standard Deviation); unit: % of area
Arm/Group | Imatinib Mesylate | Placebo
Number analyzed (Participants) | 21 | 27
% of area | 0.0002 (0.02) | 0.0002 (0.02)
Statistical Analysis 1: Comparison: Imatinib Mesylate vs Placebo; Test type: Superiority; p = 0.25, Regression, Linear; Adjusted for baseline

22. Secondary Outcome: Bronchoalveolar Lavage Histamine
Description: Change in bronchoalveolar lavage histamine levels from baseline
Time Frame: 6 months after start of treatment
Measure: Mean (Standard Deviation); unit: nM
Arm/Group | Imatinib Mesylate | Placebo
Number analyzed (Participants) | 21 | 26
nM | 2.1 (6.3) | -1.1 (13.4)
Statistical Analysis 1: Comparison: Imatinib Mesylate vs Placebo; Test type: Superiority; p = 0.54, Regression, Linear; Adjusted for baseline

23. Secondary Outcome: Urinary Prostaglandin D2
Description: Change in urinary Prostaglandin D2 levels from baseline
Time Frame: 6 months after start of treatment
Measure: Mean (Standard Deviation); unit: ng/mg Creatinine
Arm/Group | Imatinib Mesylate | Placebo
Number analyzed (Participants) | 20 | 20
ng/mg Creatinine | -0.30 (1.5) | 0.39 (1.73)
Statistical Analysis 1: Comparison: Imatinib Mesylate vs Placebo; Test type: Superiority; p = 0.18, Regression, Linear; Adjusted for baseline

24. Secondary Outcome: Bronchoalveolar Lavage Cysteinyl Leukotrienes
Description: Change in bronchoalveolar lavage cysteinyl leukotrienes levels from baseline
Time Frame: 6 months after start of treatment
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Imatinib Mesylate | Placebo
Number analyzed (Participants) | 21 | 26
pg/mL | 3.0 (37.3) | 6.5 (32.9)
Statistical Analysis 1: Comparison: Imatinib Mesylate vs Placebo; Test type: Superiority; p = 0.56, Regression, Linear; Adjusted for baseline

25. Secondary Outcome: Urinary Leukotriene E4
Description: Change in urinary leukotriene E4 levels from baseline
Time Frame: 6 months after start of treatment
Measure: Mean (Standard Deviation); unit: ng/mg Creatinine
Arm/Group | Imatinib Mesylate | Placebo
Number analyzed (Participants) | 17 | 13
ng/mg Creatinine | 0.07 (0.65) | 0.01 (0.18)
Statistical Analysis 1: Comparison: Imatinib Mesylate vs Placebo; Test type: Superiority; p = 0.47, Regression, Linear; Adjusted for baseline

26. Secondary Outcome: Change in Sputum Supernatant Differential, Supernatant Tryptase and IL-13
Description: Change in sputum eosinophil and neutrophil percentage. Change in sputum supernatant tryptase as measured by ELISA. Change in sputum IL-13 level as measured by ELISA.
Time Frame: baseline to 24 weeks
Population: Sputum sample slide preparation quality was poor and samples meeting quality control were insufficient for analysis of sputum differential.
  Insufficient study funds prevented assessment of sputum tryptase. IL-13 was below the detection limit of assay in sputum supernatant.
Arm/Group | Imatinib Mesylate | Placebo
Number analyzed (Participants) | 0 | 0

27. Secondary Outcome: Change in Inflammatory Mediators in Exhaled Breath Condensate
Description: Assessment of change in eicosanoids in the exhaled breath condensate
Time Frame: baseline to week 24
Population: The exhaled breath condensate was not processed for inflammatory mediators.
Arm/Group | Imatinib Mesylate | Placebo
Number analyzed (Participants) | 0 | 0

28. Secondary Outcome: Change in Number of Self-Reported Asthma Symptom Free Days
Time Frame: baseline to week 24
Population: Self-reported asthma symptom free days were not entered into the study database.
Arm/Group | Imatinib Mesylate | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from randomization to study drug vs. placebo up to 24 weeks.
Arm/Group | Imatinib Mesylate | Placebo
Serious Adverse Events (participants affected / at risk) | 3/32 | 5/30
Other Adverse Events (participants affected / at risk) | 29/32 | 23/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Imatinib Mesylate (N=32) | Placebo (N=30)
Asthma Exacerbation (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (6)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Leg Cramps (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Acute URI (Infections and infestations) | 0 (0) | 1 (1)
Ankle Dislocation (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Angioedemia (Immune system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Imatinib Mesylate (N=32) | Placebo (N=30)
Leukopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Fatigue (General disorders) | 0 (0) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 4 (4) | 3 (4)
Pruritis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 5 (6) | 2 (2)
Nausea/Vomiting (Gastrointestinal disorders) | 6 (7) | 2 (2)
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 9 (11) | 12 (18)
Pneumonia (Infections and infestations) | 0 (0) | 2 (2)
Urinary Tract Infection (Infections and infestations) | 2 (2) | 1 (1)
Gastroenteritis (Infections and infestations) | 2 (2) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 4 (6) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Abnormal LFTs (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Muscle Cramps (Musculoskeletal and connective tissue disorders) | 6 (10) | 1 (1)
Lightheadedness (Nervous system disorders) | 0 (0) | 2 (2)
Back/Shoulder Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Headache (Nervous system disorders) | 2 (2) | 1 (1)
Asthma Exacerbation (Respiratory, thoracic and mediastinal disorders) | 14 (16) | 13 (20)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No